CLINICAL TRIAL: NCT02834000
Title: Haemodynamic Response to General Anaesthesia Induction in Elective Orthopaedic Surgery Patients Using Non-invasive Cardiovascular Monitoring
Brief Title: Haemodynamic Response to General Anaesthesia in Healthy Orthopaedic Patients
Acronym: HRespToAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Marcela P. Vizcaychipi, Consultant in Anaesthesia and Intensive Care Medicine, Honorary Senior Clinical Lecturer, Divisional Research Lead for Planned Care Surgery and Clinical Support, Chelsea and Westminster NHS Foundation Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14/WM/0179
Record Dates: First submitted 2016-05-10; First posted 2016-07-15 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (No Intervention): We will compare the standard monitored group of patients with the LiDCO rapid™ monitored group. The control group will compose of patients supervised in a standard way.
- LiDCO rapid™ CNAP monitoring (Experimental): Young, healthy adult patients (ASA I and II) undergoing elective orthopaedic surgery under general anaesthesia will be included in to this study. We will compare the standard monitored group of patients with the LiDCO rapid™ monitored group. We will use in the LiDCO rapid™ CNAP monitoring group, the continuous real time haemodynamic monitoring through non-invasive arterial pressure waveform. The monitor LiDCO rapid™ CNAP permits, through analysis the arterial blood pressure trace, to acquire information about CO, SVR, HR variability, SV and BIS.
  Interventions: Device: LiDCO rapid™ CNAP monitoring

INTERVENTIONS:
Device: LiDCO rapid™ CNAP monitoring — LiDCO rapid™ CNAP monitoring allows through analysis of the arterial blood pressure trace to acquire information about CO, HR variability, SVR, SV and BIS during general anaesthesia.
  Other Names: http://www.lidco-ir.co.uk
  Arms: LiDCO rapid™ CNAP monitoring

SUMMARY:
Continuous cardiovascular monitoring as part of management of high-risk surgical patients is widely practiced, however its role in low-risk surgical patients is unclear. Detailed monitoring of cardiovascular parameters from pre-induction stage allows clinicians to individualise anaesthetic management in the perioperative period. The investigators' aim was to investigate haemodynamic and Bispectral Index (BIS) changes in healthy patients undergoing surgery following induction of anaesthesia with propofol using a continuous non-invasive blood pressure device (LiDCOrapid™).

DETAILED DESCRIPTION:
Recruitment Orthopaedic surgical teams, anaesthetists and theatre staff were made aware of the study that was being conducted at the investigators' institution. Prospective subjects that met the inclusion criteria were identified from the hospital operating theatre's database two weeks prior to surgery. A letter, which contained the study's objectives and methods, was sent out to all patients. Subsequently, a telephone call was made to patients one week before surgery to clarify any queries they had. Consent was obtained on the morning of surgery. All study participants provided written informed consent.

Peri-operative monitoring LiDCO™ CNAP and BIS monitoring were attached prior to induction of anaesthesia in the anaesthetic room of the operating theatre. A standardised anaesthetic technique was used for every participant, consisting of propofol induction, sevoflurane maintenance to a target BIS (40-60) and opioid analgesia with fentanyl. Participants underwent positive pressure ventilation to a tidal volume of 8ml/kg.

Measurements of the following variables were taken continuously from pre-induction to time of extubation: heart rate, mean arterial blood pressure, stroke volume, cardiac output, systemic vascular resistance and BIS. Data recorded up to 3 minutes following propofol injection was analysed to capture the post-induction period. Further measurements were taken in recovery room. The total quantity and type of fluids, drugs administered, time of tourniquet application and removal (if performed), and the duration of the operation were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the study were those aged 18-45 years undergoing elective lower limb arthroscopic procedures with an American Society of Anesthesiologists (ASA) Grade of I-II.

Exclusion Criteria:

* Patients unable or unwilling to provide valid informed consent,
* Patients undergoing regional anaesthesia,
* Patients that have contraindications to the LiDCO rapid™ CNAP monitoring (cardiac arrhythmias, aortic regurgitation and digital ischaemia) and BIS monitoring (hypersensitivity to adhesive use) and refusal of surgical, anaesthetic or operating theatre team.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Cardiac output (mls blood/ minute) | From induction up to 3 minutes

SECONDARY OUTCOMES:
Depth of anaesthesia using Bispectral Index (BIS) | From induction up to 3 minutes

IPD SHARING:
Plan to Share IPD: Yes